CLINICAL TRIAL: NCT06123936
Title: Impact on Influenza Vaccination Rates of a Telephone Text Message Recall From the Attending Physician - a Cluster Randomized, Controlled and Pragmatic Trial
Brief Title: Impact on Influenza Vaccination Rates of a Telephone Text Message Recall From the Attending Physician
Acronym: GP-FluRecall
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP220090; N° IDRCB: 2022-A00896-37 (Other: ANSM)
Record Dates: First submitted 2023-10-16; First posted 2023-11-09 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Influenza Viral Infections
Keywords: Reminder; Vaccination campaign; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): GPs selected at random in the intervention arm "Recall" will recall their patients to be vaccinated via the recall module integrated into their Eo medical software
  Interventions: Other: Reminder
- No intervention group (No Intervention): GPs in the ""usual care"" or ""control"" arm will not recall their patients to be vaccinated. GPs with their medical software.
  They will worked as usual.

INTERVENTIONS:
Other: Reminder — At mid-campaign, GPs in the interventional arm will recall their patients to be vaccinated via the reminder module Eo software
  * This recall will be carried out as follows: patients whose medical records include a number likely to receive telephone text messages will be recalled by this means Two generic messages that doctors can choose will be proposed by the call-back module integrated into the Eo medical software
  * In addition, the recall module will offer to send a postal letter with the same content as the text message to patients who do not have a mobile phone number in the business software but do have a postal address
  * The recall module will also provide the doctor with a list of patients who have neither a mobile phone number or a postal address, so that he can recall them to be vaccinated orally by landline telephone or in consultation when they next visit.
  The type of recall and the date of it will be notified in the medical file of each patient.
  Arms: Experimental group

SUMMARY:
This study is a clinical trial designed to assess the impact on influenza vaccination rates among people aged over 65 of a telephone text message recalling them to be vaccinated by their GP. Twenty-two GPs will be randomly selected in each arm (recall versus usual care, 1:1). Each GP will include a maximum of 210 patients by random selection from their patient list. A difference of 4 percentage points is expected between the two arms at the end vaccination campaign in the vaccination rate.

DETAILED DESCRIPTION:
This is an open-label trial with 2 arms: an interventional or "recall" arm and a "usual care" or control arm. Cluster randomization at the physician level was chosen to avoid contamination within the same patients group. Physicians will be randomized at the start of the vaccination campaign in one of the two arms (1:1), and all patients eligible (with a maximum of 210 per doctor) to be vaccinated will be recalled or not, depending on their GPs arm.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for physicians are:

* To be a GPs
* To be based in Ile-de-France (Paris region, France)
* To be a user of the Eo medical software

The patients inclusion criteria are:

* belonging to the list of attending physicians of the participating GPs
* being 65 years of age or older
* having a medical file in the GP's Eo medical software
* having been selected at random if the number of patients aged 65 or over exceeds 210 patients (for 44 participating GPs).

Exclusion Criteria:

* Patients for which their attending physicians considers participating inappropriate (e.g. palliative care)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 8400 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The influenza vaccination rate will be calculated as the ratio between the number of patients vaccinated (those who will report having been vaccinated in the questionnaire send at the end of the campaign) and the number of patients aged 65 years and over | 12 months
  The influenza vaccination rate will be calculated as the ratio between the number of patients vaccinated (i.e., those who will report having been vaccinated during the vaccination campaign in the questionnaire send at the end of the campaign) and the number of patients aged 65 years and over.

SECONDARY OUTCOMES:
1/ Social inequalities related to the intervention, based on individual and ecological indicators (social deprivation index for example) will be estimated via absolute indicators (SII: slope of the inequality index) and relative (RII: relative inequality | 1 year
  At the end of the vaccination campaign, the GPs will send patients a postal mail containing: an accompanying explanatory letter, the patient questionnaire, and a pre-addressed and prepaid envelope for the return of the completed questionnaire to their attending physician.
2/ Acceptability of reminders (in the intervention arm only) based on the description of the patients answers to the related question in the questionnaires. This outcome is assessed by questionnaire. | 1 year
  At the end of the vaccination campaign, the GPs will send patients a postal mail containing: an accompanying explanatory letter, the patient questionnaire, and a pre-addressed and prepaid envelope for the return of the completed questionnaire to their attending physician.
3/ Reasons for non-vaccination will be described (stratified by trial arm) based on the description of the patients answers to the related question in the questionnaires.This outcome is assessed by questionnaire. | 1 year
  Reasons for non-vaccination will be described (stratified by trial arm) based on the description of the patients answers to the related question in the questionnaires.
4/ Characteristics of participating GPs based on the description of the physicians answers to the related question in the questionnaires. These outcomes are assessed by the physician questionnaire. | 1 year
  At the beginning of the study, participating GPs will answer a short questionnaire about their main characteristics (Sex, Date of birth, Size of the patients list...).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent RIGAL, Professor, Principal Investigator — Université de Paris-Saclay
Locations (1):
- Cabinet medical Lahire (01), Paris, France

IPD SHARING:
Plan to Share IPD: No